CLINICAL TRIAL: NCT02494960
Title: Brief Tobacco Cessation Intervention: a Randomized Controlled Trial in Guangdong, China
Brief Title: Brief Tobacco Cessation Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Lam Tai-Hing, Chair Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MegaRCT
Record Dates: First submitted 2015-07-08; First posted 2015-07-10 (Estimated); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Smoking
Keywords: smoking cessation intervention
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control Group (Placebo Comparator): The doctor will offer a placebo intervention.
  Interventions: Behavioral: Placebo intervention
- Intervention Group A (Experimental): The doctor will offer the brief smoking cessation AWARD model .
  At 1-month follow-up survey, trained study personnel will repeat the brief smoking cessation AWARD model .
  Interventions: Behavioral: The brief smoking cessation AWARD model
- Intervention Group B (Experimental): The doctor will offer the brief smoking cessation AWARD model.
  Interventions: Behavioral: The brief smoking cessation AWARD model

INTERVENTIONS:
Behavioral: The brief smoking cessation AWARD model — * Ask whether or not the patient currently smokes
  * Warn the patients that at least one out of two smokers will be killed by smoking. Recent research shows that two out of three smokers will be killed by smoking. The 10-20-second script could be like 'I warn you that smoking can kill you by many serious diseases and that your chance to be killed prematurely by smoking is about 50% to 67%.
  * Advice the patients to quit now or as soon as possible because quitting can reduce the excess risks substantially.
  * Refer the patients to a smoking cessation clinic or call telephone quitlines (if available) as soon as possible, emphasizing that smoking cessation counsellors are caring and helpful.
  * Do it again: Repeat the intervention among smokers who fail to quit or relapse, and encourage them to try to quit again.
  Arms: Intervention Group A; Intervention Group B
Behavioral: Placebo intervention — Advice the smokers to eat vegetables, and engage in regular physical activities, and offer the smokers a card which contains information about the benefits of eating vegetables and a pictorial information leaflet which shows the recommended amount of vegetables and fruits an adult should eat a day
  Arms: Control Group

SUMMARY:
Traditional smoking cessation clinics and telephone quitlines are expensive and 'passive' as they require motivated smokers to visit the clinic or make a phone call to seek help. However, in most middle-resource countries, smoking cessation clinics are not well publicized. Most health care professionals (HCP) are not active in performing smoking cessation counselling to their patients. They are not aware of the available smoking cessation services or the benefits of such services and hence do not refer smokers to smoking cessation services. On the other hand, physicians play a critical role in reducing tobacco use by advising smoking patients to quit (Richmond, 1999). Physician's advice to quit smoking not only motivates smokers to quit but also increases their quitting confidence (Fiore et al., 2000; Ossip-Klein et al., 2000).

Brief smoking cessation interventions have been shown to be effective with strong evidence from randomized controlled trials (RCTs), however, it is no evidence to show that longer interventions are more effective than shorter interventions. If carried out in routine clinical practice by all physicians and other HCP, brief interventions can potentially benefit a great number of smokers and increase smoking cessation rate. Therefore, we propose to examine the effect of a brief smoking cessation counselling intervention (10-20 seconds AWARD model) among patients using a randomized controlled trail (RCT) design in Guangdong province, China

This project aims to evaluate the effect of physicians' brief smoking cessation intervention (AWARD model) in real busy clinic settings using a randomized controlled trial (RCT) design.

DETAILED DESCRIPTION:
Smokers will be recruited from the internal medicine outpatient clinics at the participating hospitals (the general nonprofit public hospitals) and community health centers. Same as the pilot study, trained doctors will ask all visiting patients during clinic consultation whether they smoke, confirm eligibility, provide information sheet and seek oral agreement to be followed up by telephone after clinic consultation. If eligible and oral consent obtained, the doctor will fill the recruitment form.

The doctors will randomly allocate the enrolled patient into intervention or control group using SNOSE method. This method will ensure allocation concealment. If the patient refuses to participate, the doctor will note on the summary form. Enrolled patients' medical records will be marked with a sticker (red for intervention group, green for control group) so they will not be recruited again if they come back to the participating hospital.

At the end of each clinic session, the doctors will immediately fill the rest part of the summary form and send the recruitment form and summary form to trained research assistants by email or WeChat. The research assistants will enter all information into a web-based or app-based study management system (SMS) using tablet PC.

For smokers in intervention group, the doctor will offer a brief (10-20 seconds) WAR smoking cessation intervention (Warn the smokers that at least one out of two smokers will be killed by smoking, and according to WHO, two out of three smokers will be killed by smoking; Advice the smokers to quit now or as soon as possible; and Refer the smokers to a smoking cessation clinic or telephone quitlines by offering a referral card which contains the contact information of the smoking cessation clinics and/or quitlines as well as a pictorial information leaflet which explains the risks of smoking). For control group, the doctor will offer a brief (10-20 seconds) placebo intervention (Advice the smokers to eat vegetables, and offer the smokers a card which contains information about the benefits of eating vegetables and a pictorial information leaflet which shows the recommended amount of vegetables and fruits an adult should eat a day).

Within 3 days after enrolment (T1), study personnel will call the participants using the tablet PC with questionnaire program to invite them to complete a short baseline survey.

At 1-month FU (T2), study personnel will call the participants using the tablet PC with questionnaire program to assess his/her smoking and quitting outcomes. After the assessment, trained study personnel will get the information about the participants' group status from the tablet PC. For Group C, the trained study personnel will end the phone call without further assessment or intervention. For Group I, the trained study personnel will use the tablet PC to randomly assign the participant to Group I-A or I-B.

For Group I-A, trained study personnel will repeat the brief (10-20 seconds) AWARD intervention (Warn the smokers that at least one out of two smokers will be killed by smoking, and according to WHO, two out of three smokers will be killed by smoking; Advice the smokers to quit now or as soon as possible; and Refer the smokers to a smoking cessation clinic or telephone quitlines by offering the contact information of the smoking cessation clinics and/or quitlines); for Group I-B, trained study personnel will end the phone call without further questions or actions.

At 3-month FU (T3), study personnel will use the programmed tablet PC to call participants and measure his/her smoking patterns and quitting efforts.

At 6- and 12-month FU (T4&T5), study personnel will use the programmed tablet PC to call participants and measure his/her smoking patterns and quitting efforts again. Participants who report that they have been abstained from nicotine for ≥7 days will be invited to complete biochemical validation in clinics. Exhaled CO less than 4ppm and salivary cotinine less than 10ng/ml tested by NicAlert® strips (www.nymox.com) will be treated as validated abstinence. If for any reason, the participants are not able to complete the biochemical validation, study personnel will use the programmed tablet PC to conduct a non-biochemical validation survey to validate whether or not the participants have been abstained from nicotine.

Study personnel will always be blinded to participants' group status at follow-up interviews (single blinded). Subjects will be randomly allocated to study personnel for follow-up interviews, so subjects are likely to be interviewed by different study personnel in this study.

T-test will be conducted to compare the primary (a) outcomes and the secondary outcomes. Separate multivariate logistic regression model will be performed for each of the three groups (i.e., I-A, I-B, and C) between the baseline and the 12-month follow-up, controlling for age, gender, education, and income to determine whether the outcome of interests (quitting rate and smoking reduction rate) had increased, remained unchanged, or decreased. Change (e.g., increase or decrease) will be considered significant if p <.05.

Multivariate logistic regression models will also be used to examine if the smoking cessation intervention is associated with successful quitting and smoking reduction, as well as other factors (e.g., demographic variables) associated with successful quitting and smoking reduction.

Sensitivity test based on the result of physicians' fidelity check will be conducted to determine the effect of the physician's very brief smoking cessation counselling on quitting and smoking pattern changes. The fidelity check will evaluate the adherence of physicians' implementation to the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients aged 18 years or above
* Smoke on at least 1 day in the past 30 days
* Chinese residents able to communicate in Chinese (Mandarin or Cantonese)
* Has a telephone

Exclusion Criteria:

* Smokers currently receiving smoking cessation interventions
* Smokers currently enrolled in other smoking cessation trials
* Smokers who need special care on quitting and are not suitable for AWARD intervention (determined by his/her doctor)
* Smokers with communication difficulties (physical or cognitive condition)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13671 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Smokers' self-reported 7-day point prevalence quitting rate | up to 12-months follow-up
  Self-reported tobacco abstinence in the past 7 days

SECONDARY OUTCOMES:
Biochemically validated quit rate | 6- and 12-months follow-up
  Tobacco abstinence validated by exhaled carbon monoxide (<4ppm) and saliva cotinine (<10ng/ml)
Non-biochemically validated quit rate | 6- and 12-months follow-up
  Tobacco abstinence verified by the interviewers
Self-reported sustained nicotine abstinence | 1- and 3-month follow-up
  Self-reported tobacco abstinence in the past 30 days
Smoking reduction (cigarette or other tobacco product use decreased by at least 50%) among continuing smokers | 1-, 3-, 6- and 12-months
  Smoking reduction (cigarette or other tobacco product use decreased by at least 50% compared with baseline) among continuing smokers
Number of quit attempts | 1-, 3-, 6- and 12-months
  Self-reported intentionally no smoking for at least 24 hours
Proportion of smokers visit smoking cessation clinics or call the telephone quitlines | 1-, 3-, 6- and 12-months
  Proportion of smokers visit smoking cessation clinics or call the telephone
Body weight | 1-, 3-, 6- and 12-month FU
  Body weight

CONTACTS AND LOCATIONS:
Overall Officials: Tai hing Lam, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- 5/F William MW Mong Block, LKS Faculty of Medicine Building, 21 Sassoon Road, Pokfulam, Hong Kong, Guangdong, China